CLINICAL TRIAL: NCT06729931
Title: Quantitative C-Reactive Protein for Differentiation Between Tuberculous and Malignant Pleural Effusion: an Institutional Cross-Sectional Study
Brief Title: Quantitative C-Reactive Protein for Differentiating Tuberculous and Malignant Pleural Effusion: a Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Asim Shrestha, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 225(6-11)E2079/080
Record Dates: First submitted 2024-12-07; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pleural Effusion; Malignant Pleural Effusions; Tuberculous Pleural Effusion
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tuberculous Pleural Effusion: Patients diagnosed with tuberculous pleural effusion based on pleural fluid ADA, AFB/GeneXpert, or pleural/lung tissue biopsy.
  Interventions: Diagnostic Test: Pleural Fluid Quantitative C-Reactive Protein (Q-CRP) Measurement
- Malignant Pleural Effusion: Patients diagnosed with malignant pleural effusion through pleural fluid cytology or pleural/lung tissue biopsy, supported by radiological findings.
  Interventions: Diagnostic Test: Pleural Fluid Quantitative C-Reactive Protein (Q-CRP) Measurement

INTERVENTIONS:
Diagnostic Test: Pleural Fluid Quantitative C-Reactive Protein (Q-CRP) Measurement — The intervention involves the measurement of Quantitative C-Reactive Protein (Q-CRP) levels in pleural fluid obtained from patients presenting with lymphocytic exudative pleural effusion. The Q-CRP test is performed using standardized laboratory methods to quantitatively analyze CRP levels, which are then compared between patients with confirmed tuberculous pleural effusion and those with malignant pleural effusion. This diagnostic approach aims to evaluate the efficacy of pleural fluid Q-CRP as a biomarker to differentiate between these two conditions. No therapeutic or invasive interventions are introduced as part of this study beyond routine diagnostic procedures.
  Other Names: Pleural Fluid CRP; Quantitative CRP Analysis

SUMMARY:
The goal of this observational study is to evaluate the role of pleural fluid Quantitative C-Reactive Protein (Q-CRP) levels in distinguishing between tuberculous and malignant pleural effusion in adult patients with lymphocytic exudative pleural effusion.

The main questions it aims to answer are:

Is pleural fluid Q-CRP significantly higher in tuberculous pleural effusion compared to malignant pleural effusion? What is the optimal cutoff value of pleural fluid Q-CRP to differentiate between these conditions?

Participants will:

Undergo diagnostic procedures such as pleural fluid analysis, including ADA and cytology.

Provide pleural fluid samples for Q-CRP measurement. Have additional diagnostic imaging or biopsies if clinically indicated.

Researchers will compare Q-CRP levels between the tuberculous pleural effusion group and the malignant pleural effusion group to determine its diagnostic accuracy, including sensitivity, specificity, and predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Patients presenting with lymphocytic exudative pleural effusion confirmed by Light's criteria.
* Lymphocyte predominance in pleural fluid (≥ 50% of differential count).

Exclusion Criteria:

* Patients who refuse to provide consent for study participation.
* Patients requiring biopsy under general anesthesia but found unfit for the procedure.
* Non-tuberculous and non-malignant lymphocytic exudative pleural effusions identified during diagnostic evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and above who presented with lymphocytic exudative pleural effusion at the Thoracic Surgery Unit, Department of CTVS, MCVTC, and the Department of Pulmonology, TUTH, Kathmandu, Nepal. Participants were recruited based on specific inclusion and exclusion criteria. Diagnostic evaluations, including pleural fluid analysis and additional testing (e.g., ADA, AFB, GeneXpert, cytology, or biopsy), were conducted to classify cases as tuberculous or malignant pleural effusion. Only confirmed cases of these conditions were included in the final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Comparison of Pleural Fluid Quantitative C-Reactive Protein (Q-CRP) Levels Between Tuberculous and Malignant Pleural Effusion | Within 1 year (from November 2022 to October 2023)
  The primary outcome is the difference in pleural fluid Quantitative C-Reactive Protein (Q-CRP) levels between patients diagnosed with tuberculous pleural effusion and those with malignant pleural effusion. The study evaluates the diagnostic utility of Q-CRP levels as a biomarker by comparing mean values, sensitivity, specificity, and Area Under the Receiver Operating Characteristic (ROC) curve for differentiation between the two conditions.

SECONDARY OUTCOMES:
Sensitivity and Specificity of Pleural Fluid Q-CRP Cut-off Values for Differentiating Tuberculous and Malignant Pleural Effusion | Within 1 year (from November 2022 to October 2023)
  The secondary outcome evaluates the diagnostic performance of pleural fluid Q-CRP cut-off levels derived from the ROC curve analysis. Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) are calculated to assess the utility of Q-CRP in accurately differentiating tuberculous pleural effusion from malignant pleural effusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medicine, Maharajgunj, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request for research purposes following publication of the study results